CLINICAL TRIAL: NCT06107283
Title: Study of the Reduction of the Prescriptions of Benzodiazepines and Related After the Discharge of a Service of Follow-up Care and Geriatric Rehabilitation
Brief Title: Study of the Reduction of the Prescriptions of Benzodiazepines and Related
Acronym: BZD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8787
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Depression in Old Age
Keywords: Depression in Old Age; Benzodiazepines drugs; Geriatrics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The significant consumption of Benzodiazepines and related drugs in the elderly outside of good practice recommendations is a major issue in the care of the elderly. Adverse effects have been the subject of numerous studies, leading to falls, addictions and even deaths. The general practitioner is often faced with long-term medication intake which is not consistent with a good benefit/risk balance, but stopping or reducing the dosage remains a problem in current practice.

The Aftercare and Geriatric Rehabilitation services due to their operation (several weeks of hospitalization) seek to adapt the patient's therapies in order to obtain the most convincing benefit/risk balance possible. A reduction or withdrawal of treatments with Benzodiazepines or related drugs are therefore frequently initiated.

DETAILED DESCRIPTION:
The aim of this research is to quantify among the patients who benefited from a dosage reduction of Benzodiazepines and related drugs during a stay in the Geriatric Care and Aftercare and Rehabilitation department, the number of patients who had an increase of this treatment within 12 weeks following discharge from hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 75 years old)
* Subject discharged from a geriatric Follow-up Care and Rehabilitation service for whom a reduction in the dosage of Benzodiazepines and related drugs was carried out during hospitalization and who returned home (individual or EHPAD) after hospitalization.
* Subject not opposing, after information, the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study.
* Subject having treatment with Benzodiazepine to prevent recurrence of epileptic seizures.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Major subject (≥ 75 years old) discharged from a geriatric Follow-up Care and Rehabilitation service for whom a reduction in the dosage of Benzodiazepines and related drugs was carried out during hospitalization and who returned home (individual or EHPAD) after hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
The number of patients who had an increase in Benzodiazepines in the 12 weeks following discharge from hospitalization. | 12 weeks following discharge from hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Gériatrie - Service de Soins de Soins Médicaux et de Réadaptation - CHU de Strasbourg - France, Strasbourg, France